CLINICAL TRIAL: NCT00774553
Title: A Randomized, Single-Blind, Placebo-Controlled, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Multiple Ascending Oral Doses of AZD1656 in Subjects With T2DM Treated With Metformin
Brief Title: To Evaluate Safety and Tolerability After Multiple Oral Doses of AZD1656 in Type 2 Diabetes Patients on Top of Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1020C00015
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Dose titration of oral suspension to a tolerable dose given twice daily for 10 days.
  Arms: 1
Drug: Placebo — Dose titration of oral suspension to a tolerable dose given twice daily for 10 days.
  Arms: 2

SUMMARY:
The purpose of this study is to assess safety and tolerablility of AZD1656 after multiple repeated oral doses in patients with type 2 diabetes on top of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (with non child-bearing potential)
* Diagnosed diabetes Mellitus patients treated with metformin alone or one other anti-diabetic drugs. Stable blood sugar control indicated by no changed treatment within 3 months prior to study start.t
* HbA1c <11 % at screening (HbA1c value according to international DCCT standard)

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within two weeks before the first administration of the IP
* History of ischemic heart disease, stroke, transitorisk ischemic attack or symptomatic peripheral vascular disease
* Clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety variables (AE, BP, pulse, plasma glucose, laboratory variables, weight and ECG) | Blood samples taken repeatedly during 24 hours on study day sessions

SECONDARY OUTCOMES:
Pharmacokinetic variables | Blood samples taken repeatedly during 24 hours on study day sessions
Pharmacodynamic variables | Blood samples taken repeatedly during 24 hours on study day sessions

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof.,, Study Director — AstraZeneca R&D Mölndal; Dr Emanuel DeNoia, MD, Principal Investigator — Healthcare Discoveries LLC Icon Development Solutions; Sanjay Sharma, MD, Principal Investigator — Veeda Clinical Research Pvt. Ltd
Locations (2):
- Research Site, San Antonio, Texas, United States
- Research site, Ahmedabad, India